CLINICAL TRIAL: NCT06159868
Title: Physiotherapy and Optimised Enteral Nutrition In the Post-acute Phase of Critical Illness (PHOENIX): A Randomised Controlled Feasibility Trial
Brief Title: Physiotherapy and Optimised Nutrition in Survivors of Critical Illness
Acronym: PHOENIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DM633323
Record Dates: First submitted 2023-11-28; First posted 2023-12-07 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Critical Illness
Keywords: physiotherapy; nutrition; rehabilitation; intensive care; exercise
MeSH Terms: conditions — Critical Illness; Motor Activity | interventions — Rehabilitation; Standard of Care

STUDY DESIGN:
Intervention Model Description: A mixed-methods, multicentre, randomised controlled feasibility study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study outcome assessors will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Structured and individualised physiotherapy in combination with optimised nutrition delivered by s specialist critical care rehabilitation team
  Interventions: Other: Structured physiotherapy and rehabilitation
- Control (Active Comparator): Standard ward based care
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Structured physiotherapy and rehabilitation — Comprehensive baseline assessment of function and nutrition using indirect calorimetry to identify nutritional requirements, to create and individualised plan for followed by daily targeted mobility retraining, exercise and nutrition.
  Arms: Intervention
Other: Standard care — Standard ward based care provided by usual care teams
  Arms: Control

SUMMARY:
The goal of this randomised controlled feasibility study is to assess the feasibility and acceptability of individualised physiotherapy and optimised nutrition, delivered on the ward following discharge from intensive care to increase days alive and out of hospital, as well as the proposed methodology to optimise design and delivery for a definitive evaluation trial. Specific objectives are:

i. To assess acceptability of the intervention to users and providers. ii. To assess feasibility of recruitment procedures for a future trial. iii. To estimate recruitment, retention and measure completion rates for a future trial.

Participants will receive a combination of structured, individualised physiotherapy and optimised nutrition, beginning immediately following recruitment and continuing for up to 14days or hospital discharge, whichever is sooner. As a feasibility trial the primary outcomes to be assessed are around study feasibility. The investigators will also compare clinical outcomes for the intervention participants in comparison to those receiving standard care to see if the intervention increases the number of days alive and out of hospital within 30 days of recruitment.

DETAILED DESCRIPTION:
Research question Is it feasible and acceptable to undertake a randomised controlled trial evaluating the clinical and cost-effectiveness of an individualised physiotherapy and nutrition support intervention, delivered on the ward following ICU discharge, in adult survivors of critical illness?

Background Each year in the UK, 140,000 patients are discharged from intensive care units (ICU) to general hospital wards, almost all with complex rehabilitation needs. Eighty-four percent of patients still require nutritional support and 98% are not physically independent. Despite this, many are discharged from ICU without a nutrition plan and failure to recognise malnutrition is common. Consequently, malnutrition persists in the ward environment, leading to poor outcomes in itself, and additionally acts as a barrier to successful physical rehabilitation. This transition from intensive care to the ward represents a key stage in the recovery journey, and a window for optimising physical independence prior to hospital discharge, decreasing the need for support in the community. However, uncertainty as to how best to provide ongoing rehabilitation combining adequate nutrition and exercise on the general ward has driven widespread variation in practice.

The investigators have previously shown the benefits of delivering a structured rehabilitation strategy in the ICU. However, the ward environment poses different challenges to the development of an integrated rehabilitation pathway. There is a need to evaluate the clinical and cost-effectiveness of structured rehabilitation strategies when delivered outside the ICU.

Aims To evaluate the feasibility and acceptability of conducting a randomised controlled trial evaluating the clinical and cost-effectiveness of structured, individualised physiotherapy and nutritional support in ward-based patients following ICU discharge.

Objectives:

i. To assess acceptability of the intervention to users and providers ii. To assess feasibility of recruitment procedures for a future trial iii. To estimate recruitment, retention and measure completion rates

Methods PHOENIX is a two-centre, allocation-concealed, open-label, parallel group, randomised controlled feasibility trial with integrated qualitative evaluation of acceptability.

The investigators will recruit sixty adult survivors from intensive care units at two university hospitals, with ongoing physiotherapy and nutritional needs at ICU discharge. Participants will be randomised on a 1:1 basis to receive the structured rehabilitation intervention or standard care. The intervention comprises enhanced physiotherapy, delivered by a specialist critical care team, in combination with optimised nutrition guided by indirect calorimetry.

Primary feasibility outcomes are recruitment and retention rates, and intervention fidelity. Acceptability will be evaluated through semi structured interviews of participants and staff.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years) that received ≥ 4 days advanced respiratory support (defined as invasive or non-invasive ventilation) on ICU,
* Alive at ICU discharge
* On-going physiotherapy and dietetic rehabilitation needs identified by the PICUPS tool (Defined as patients who are unable to transfer from bed to chair independently AND not able to meet nutritional requirements independently).

Exclusion Criteria:

* Death expected within the next 72 hours,
* Poor pre-ICU admission mobility (inability to walk > 10 metres with or without an aid)
* mobilisation contraindicated (e.g., spinal injury),
* Contraindication to or inability to tolerate enteral nutrition,
* Significant brain injury and not recovered to a GCS of ≥ 14 by ICU discharge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-02-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | At recruitment within the 6 month screening window
  Proportion of patients agreeing to take part out of all those invited (recruitment rate)
Retention rate | from recruitment up to 30 days
  Proportion of participants who complete the primary outcome (retention rate)
Intervention adherence | For 14 days following recruitment
  Percentage of intervention sessions completed

SECONDARY OUTCOMES:
Days alive and out of hospital in 30 days | 30 days following recruitment
  To evaluate the number of days alive and out of hospital within the 30 days following recruitment
Physical Function | At baseline, 14 days and 30 days
  Assessed using the 30 second sit to stand test
Functional independence | At baseline, 14 days and 30 days
  Assessed using the Barthel Index
Health Related Quality of Life | At 30 days following recruitment
  Assessed using the EQ5D-5L

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University Hospitals Coventry & Warwickshire, Coventry, Midlands
  - Oxford University Hospitals Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McWilliams D, Gustafson O, Wyer N, Couper K, Kimani P, Kandiyali R, Barghouthy D, Haylett R, Richardson H, Negus-Fancey M, King E, Gallie L, Puthucheary Z. Physiotherapy and Optimised Enteral Nutrition In the post-acute phase of critical illness (PHOENIX): protocol for a mixed methods feasibility randomised controlled trial. BMJ Open. 2025 Mar 27;15(3):e100803. doi: 10.1136/bmjopen-2025-100803. PMID 40147993